CLINICAL TRIAL: NCT04643457
Title: A Phase I/IIA, Randomized, Placebo-Controlled, Single-Ascending Dose (Part A, Participant- and Investigator-Blind) and Repeated-Dose (Part B, Participant-, Investigator-, and Sponsor-Blind) Study to Investigate the Safety, Pharmacokinetics, and Efficacy of UCB9741 in Healthy Study Participants (Part A) and in Study Participants With Moderate-to-Severe Atopic Dermatitis (Part B)
Brief Title: A Study to Test the Safety, Pharmacokinetics, and Efficacy of UCB9741 in Healthy Study Participants and in Study Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0089; 2020-003639-41 (EudraCT Number)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Healthy Participants; UCB9741
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: Intravenous UCB9741 arm 1 (Experimental): Subjects randomized to this arm will receive a pre-specified single intravenous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Intravenous UCB9741 arm 2 (Experimental): Subjects randomized to this arm will receive a pre-specified single intravenous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Intravenous UCB9741 arm 3 (Experimental): Subjects randomized to this arm will receive a pre-specified single intravenous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Intravenous UCB9741 arm 4 (Experimental): Subjects randomized to this arm will receive a pre-specified single intravenous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Intravenous UCB9741 arm 5 (Experimental): Subjects randomized to this arm will receive a pre-specified single intravenous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Subcutaneous UCB9741 arm 1 (Experimental): Subjects randomized to this arm will receive a pre-specified single subcutaneous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Subcutaneous UCB9741 arm 2 (Experimental): Subjects randomized to this arm will receive a pre-specified single subcutaneous dose of UCB9741.
  Interventions: Drug: UCB9741
- Part A: Intravenous Placebo arm (Placebo Comparator): Subjects randomized to this arm will receive intravenous Placebo to maintain the blinding.
  Interventions: Drug: Intravenous Placebo
- Part A: Subcutaneous Placebo arm (Placebo Comparator): Subjects randomized to this arm will receive subcutaneous Placebo to maintain the blinding.
  Interventions: Drug: Subcutaneous Placebo
- Part B: Intravenous UCB9741 arm (Experimental): Subjects randomized to this arm will receive pre-specified intravenous doses of UCB9741.
  Interventions: Drug: UCB9741
- Part B: Intravenous Placebo arm (Placebo Comparator): Subjects randomized to this arm will receive intravenous Placebo to maintain the blinding.
  Interventions: Drug: Intravenous Placebo

INTERVENTIONS:
Drug: UCB9741 — - Pharmaceutical form: Solution Participants will receive UCB9741 during the Treatment Period.
  Arms: Part A: Intravenous UCB9741 arm 1; Part A: Intravenous UCB9741 arm 2; Part A: Intravenous UCB9741 arm 3; Part A: Intravenous UCB9741 arm 4; Part A: Intravenous UCB9741 arm 5; Part A: Subcutaneous UCB9741 arm 1; Part A: Subcutaneous UCB9741 arm 2; Part B: Intravenous UCB9741 arm
Drug: Intravenous Placebo — - Pharmaceutical form: Solution Participants will receive Placebo to maintain the blinding during the Treatment Period.
  Arms: Part A: Intravenous Placebo arm; Part B: Intravenous Placebo arm
Drug: Subcutaneous Placebo — Pharmaceutical form: Solution Participants will receive subcutaneous Placebo to maintain the blinding during the Treatment Period.
  Arms: Part A: Subcutaneous Placebo arm

SUMMARY:
The purpose of the study is to investigate the safety and tolerability of single-ascending doses of UCB9741 administered by intravenous infusion or subcutaneous injection to healthy study participants and following repeat dosing at a single dose level in study participants with atopic dermatitis. Furthermore, the clinical efficacy outcome in study participants with atopic dermatitis after administration of UCB9741 by intravenous infusion will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Participant must be 18 to 55 years of age inclusive at the time of signing the informed consent form (ICF)
* Participant must be overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant has a body mass index (BMI) within the range 18 to 30 kg/m^2 (inclusive)
* Participant can be male or female

  * A male participant must agree to use contraception during the Treatment Period and for at least 90 days after the final dose of investigational medicinal product (IMP), and refrain from donating sperm during this period
  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 90 days after the final dose of IMP

Part B:

* Participant must be 18 to 65 years of age inclusive at the time of signing the ICF
* Participant has a documented history of moderate or severe atopic dermatitis (AtD) that has been present for at least 12 months prior to initiating the study (signing of the ICF) and with:

  * validated Investigator Global Assessment (vIGA) score ≥3 at Screening (Visit 1) and Baseline (Visit 2)
  * Eczema Area and Severity Index (EASI) score of ≥14 at Screening (Visit 1) and ≥16 at Baseline (Visit 2)
  * Pruritus Numerical Rating Scale (NRS) score ≥ 3 at Screening (Visit 1) and Baseline (Visit 2)
  * ≥10% body surface area (BSA) of AtD involvement at Screening (Visit 1) and Baseline (Visit 2)
  * Either documented recent history (within 6 months before the Screening Visit) of inadequate response to treatment with topical medications (regular use of topical corticosteroids [TCS] or topical calcineurin inhibitors [TCIs]) or when topical treatments are confirmed to be otherwise medically inadvisable (eg, because of important side effects or safety risks). Inadequate response is defined as failure to achieve and maintain remission or low disease remission or a low disease activity state (validated Investigator Global Assessment (vIGA) 0=clear to vIGA 2=mild) despite treatment with a daily regimen of TCS of medium to higher potency (±TCI as appropriate), applied for at least 4 weeks or for the maximum duration recommended by the product prescribing information (eg, 2 weeks for high potency TCS), whichever is shorter
* Participant has a body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive)
* Participant can be male or female
* A male participant must agree to use contraception during the Treatment Period and for at least 60 days after the final dose of IMP, and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 60 days after the final dose of IMP

Exclusion Criteria:

Part A:

* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) or other biologic drugs as stated in this protocol
* Participant has a significant allergy to humanized monoclonal antibodies (mAbs)
* Participant has clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions
* Participant has abnormal blood pressure (BP) (outside the normal range) in a supine position after 5 minutes rest
* Participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Participant has a recent history or currently active clinically-significant bacterial, fungal, endoparasite, or viral (including hospitalization for coronavirus disease 2019 (COVID-19)) infection (within 6 months of the Screening Visit)
* Participant has a history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* Participant has a history of diabetes
* Participant has a corrected QT interval (QTc) >450 msec
* Participant has received any prescription or nonprescription medicines, including over the counter remedies and herbal and dietary supplements (other than vitamins within recommended daily dose limits), within 14 days (or 5 half-lives of the respective drug, whichever is longer) prior to the Baseline Visit, other than contraceptives (oral, implants, or intrauterine devices) or occasional use of analgesics, such as paracetamol (acetaminophen, with or without caffeine, with a maximal dose of 4 g/day and 10 g/14 days)
* Participant has received Bacillus Calmette-Guerin vaccinations within 1 year prior to the Baseline Visit or within 90 days after the final dose of IMP
* Participant has been treated with biologic agents (such as mAbs, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the Baseline Visit
* Participant has participated in another study of an IMP within the previous 90 days or 5 half-lives of the IMP (whichever longer), or is currently participating in another study of an IMP
* Participant has sensitivity to heparin or heparin-induced thrombocytopenia

Part B:

* Participant has a known hypersensitivity to any components of the IMP or other biologic drugs as stated in this protocol
* Participant has significant allergies to humanized mAbs
* Participant has clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear Immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Participant has abnormal BP (outside the normal range) in a supine position after 5 minutes rest
* Participant has ALT, AST, or ALP >1.5xULN
* Participant has a recent history of or clinically active clinically-significant, as judged by the Investigator, bacterial, fungal, endoparasite, or viral (or any history of hospitalization for COVID-19) infection (within 6 months of the Screening Visit)
* Participant has a history of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* Participant has a history of diabetes that is not well controlled with diet
* Participant has a mean QT interval (QTc) >450 msec for male study participants or >470 msec for female study participants
* Participant has received any prescription or nonprescription medicines, including over the counter remedies and herbal and dietary supplements (other than vitamins within recommended daily dose limits) within 14 days (or 5 half-lives of the respective drug, whichever is longer) prior to the Baseline Visit, other than contraceptives (oral, implants, or intrauterine devices) or occasional use of analgesics such as paracetamol (acetaminophen, with or without caffeine, with a maximal dose of 4 g/day and 10 g/14 days) or intranasal corticosteroids for seasonal rhinitis or inhaled bronchodilators and low dose inhaled corticosteroids for mild asthma
* Participant has received Bacillus Calmette-Guerin vaccinations within 1 year prior to the Baseline Visit or is anticipated to do so within 60 days after the final dose of IMP
* Participant has been treated with biologic agents (such as mAbs, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the Baseline Visit
* Participant has participated in another study of an IMP within the previous 30 days or 5 half-lives of IMP (whichever longer) from the Baseline Visit or is currently participating in another study of an IMP
* Participant has sensitivity to heparin or heparin-induced thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Incidents of treatment-emergent adverse events (TEAEs) during Part A | From Baseline up to the End of Study Visit (Week 12)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Incidents of treatment-emergent serious adverse events (TESAEs) during Part A | From Baseline up to the End of Study Visit (Week 12)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidents of TEAEs during Part B | From Baseline up to the End of Study Visit (Week 18)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Incidents of TESAEs during Part B | From Baseline up to the End of Study Visit (Week 18)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
≥75% improvement vs Baseline in Eczema Area and Severity Index (EASI75) score during Part B | Baseline, Week 12
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.

SECONDARY OUTCOMES:
Cmax from Baseline through the End of Study (EoT) Visit of Part A | From Baseline through the End Of Study Visit (Week 12)
  Cmax: Maximum observed serum concentration
Tmax from Baseline through the End of Study (EoT) Visit of Part A | From Baseline through the End of Study Visit (Week 12)
  tmax: Time to maximum observed serum concentration
AUC(0-t) from Baseline through the End of Study (EoT) Visit of Part A | From Baseline through the End of Study Visit (Week 12)
  AUC(0-t): Area under the serum concentration-time curve from time zero to time t
AUC from Baseline through the End of Study (EoT) Visit of Part A | From Baseline through the End of Study Visit (Week 12)
  AUC: Area under the serum concentration-time curve from time 0 to last observed quantifiable concentration
F% from Baseline through the End of Study (EoT) Visit of Part A | From Baseline through the End of Study Visit (Week 12)
  F%= Bioavailability of subcutaneous route
Percent change from Baseline in the Eczema Area and Severity Index (EASI) score at Week 12 of Part B | Baseline, Week 12
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
≥50% improvement vs Baseline in EASI score (EASI50) at Week 12 during Part B | Baseline, Week 12
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
≥90% improvement vs Baseline in EASI score (EASI90) at Week 12 during Part B | Baseline, Week 12
  The Eczema Area and Severity Index (EASI) is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  A participant's EASI is scored through evaluation of 4 body regions: Head and neck; Trunk; Upper extremities; Lower extremities
  The severity of disease is evaluated by assessing each of 4 clinical signs for each area:
  Erythema; Edema/papulation; Excoriation; Lichenification The severity of each clinical sign is scored as: 0=None, 1=Mild, 2=Moderate, 3=Severe.
Cmax after the final dose of Part B | Week 12
  Cmax: Maximum observed serum concentration
Tmax after the final dose of Part B | Week 12
  tmax: Time to maximum observed serum concentration
AUCtau at Week 12 of Part B | Week 12
  AUCtau: Area under the curve for the dosing interval after the final dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (10):
- Bulgaria (3):
  - Up0089 303, Pleven
  - Up0089 301, Sofia
  - Up0089 304, Sofia
- Germany (3):
  - Up0089 407, Berlin
  - Up0089 408, Heidelberg
  - Up0089 410, Leipzig
- Up0089 201, Leiden, Netherlands
- United Kingdom (3):
  - Up0089 104, Liverpool
  - Up0089 101, London
  - Up0089 103, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org